CLINICAL TRIAL: NCT01739725
Title: A Prospective Multicenter Clinical Trial to Evaluate the Comfort of the Percuflex Helical Ureteral Stent
Brief Title: Study Evaluating the Helical Ureteral Stent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Ben Chew, MD, Associate Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H11-03073
Record Dates: First submitted 2012-11-29; First posted 2012-12-03 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Kidney Calculi
Keywords: kidney stones, ureteral stent, pain,
MeSH Terms: conditions — Kidney Calculi; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Helical stent insertion (Experimental): Study participants will receive the helical stent
  Interventions: Device: Stent insertion

INTERVENTIONS:
Device: Stent insertion — The patient will receive the helical stent

SUMMARY:
The Boston Scientific Helical Stent is a unique stent designed to improve flexibility and comfort. It is designed to conform more to the shape of the ureter (hollow tube connecting the kidney and the bladder) to ultimately improve patient comfort and decrease the need for painkillers.

DETAILED DESCRIPTION:
Ureteral stents have been used for many years for a variety of clinical indications. Many surgeons routinely use ureteral stents after the endourologic removal of stones to facilitate in urine passage and facilitate excretion of any left over stones. There is a multitude of literature that reveals that most patients find ureteral stents to be uncomfortable. This discomfort often causes pain severe enough that patients anxiously anticipate stent removal, and often request early stent removal, and/or require use of pain medications that have many side effects and cause further discomfort to these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female; female patients must be sterile, post-menopausal or willing to use birth control during the course of the study
2. 19 years of age and older
3. Having undergone Shockwave Lithotripsy-SWL, or a diagnostic ureteroscopy or uncomplicated ureteroscopy for stone removal requiring retrograde placement of a ureteral stent for an anticipated duration of between 2 and 21 days
4. Willing to sign the Informed Consent Form
5. Able to read, understand, and complete patient questionnaires

Exclusion Criteria:

1. Active, symptomatic urinary tract infection
2. Non-stone related distal ureteral obstruction or stricture
3. Clinically significant trauma or significant retained stone burden that could significantly contribute to patient discomfort
4. Ureteral perforation or trauma
5. History of bladder reconstruction or interstitial cystitis
6. Spinal cord injuries

6. Pregnant or lactating females 7. Non-stone related voiding dysfunction requiring supplemental bladder drainage tubes for more than 24 hours post operatively 8. Patients with a solitary kidney 9. Chronic use of pain or anti-spasmodic medication for symptoms other than stone related pain 10. If in the opinion of the Investigator, the patient is not a suitable study candidate.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Percent of patients who have pain during the stent indwell period | 1-2 weeks
  The primary objective is to decrease the percent of patients who have pain during the stent indwell period beyond protocol-defined postoperative pain therapy from 25% for standard stents (the Control Stent in previous studies) to 10% for the Helical Stent. The previous clinical trial found that patients with Percuflex Plus stents had pain 25.2% of the time following stent insertion (J Urol 183:1037, 2010).

SECONDARY OUTCOMES:
Percent of patients requesting intervention during the stent indwell period | 1-2 weeks
  The secondary objective is to decrease the percent of patients requesting intervention during the stent indwell period.
  Interventions are defined as the following actions taken due to pain:
  1. Unscheduled Clinic visit, or
  2. Change in Pain Medication, or
  3. Early Stent Removal

CONTACTS AND LOCATIONS:
Overall Officials: Ben Chew, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No